CLINICAL TRIAL: NCT07082244
Title: Phenotype Modification Via Guided Bone Regeneration and Acellular Dermal Matrix Simultaneous to Delayed Implant Placement: A Double Arm Randomized Controlled Clinical Trial.
Brief Title: Implant Phenotype Modification Via GBR and ADM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Muhammad Saleh, Clinical Assistant Professor of Dentistry, Department of Periodotnics and Oral Medicine, School of Dentistry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00262601
Record Dates: First submitted 2025-06-04; First posted 2025-07-24 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-06

CONDITIONS: Horizontal Ridge Deficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guided bone regeneration (Active Comparator): Guided bone regeneration with collagen membrane
  Interventions: Procedure: Dental implant placement; Procedure: Guided bone regeneration with collagen membrane
- Guided bone regeneration with Phenotype modification. (Experimental): Guided bone regeneration with an allogenic dermal matrix
  Interventions: Procedure: Dental implant placement; Procedure: Guided bone regeneration with acellular dermal matrix.

INTERVENTIONS:
Procedure: Dental implant placement — Participants will have a dental implant placed at a toothless site
Procedure: Guided bone regeneration with collagen membrane — Participants will receive guided bone regeneration at a toothless site with bone substitute and a collagen membrane.
  Arms: Guided bone regeneration
Procedure: Guided bone regeneration with acellular dermal matrix. — Participants will receive guided bone regeneration at a toothless site with bone substitute and an acellular dermal matrix.
  Arms: Guided bone regeneration with Phenotype modification.

SUMMARY:
Single implant sites with bone loss can often be managed by bone grafting alone. The purpose of this study is to determine whether putting a soft tissue graft substitute over the bone graft will provide an increased benefit for improving the health, appearance, and stability of the bone and gums surrounding the implant.

DETAILED DESCRIPTION:
The study will treat patients that need a single implant at a previously edentulous site (>3 months post extraction) that requires phenotypic modification. These patients will receive an implant with simultaneous GBR, with half of the participants also receiving an ADM graft.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Subjects with a physical status of systemically healthy or suffering from mild to moderate, but well-controlled disease; American Society of Anesthesiology (ASA) I or II.
* Subjects must have one edentulous region, with at least 3 months of healing post-extraction, in the esthetic zone of the maxilla or the premolar and canine region of the mandible. This region includes the maxillary premolars, canines, and incisors.
* Subjects must have a full mouth plaque and bleeding score of less than or equal to 20%, measured at four sites per tooth.
* The patients should have a thin periodontal phenotype; bucco-lingual ridge thickness greater than 6mm.
* Seibert class I deficiency (Seibert, 1983)
* Patients willing to sign the informed consent.

Exclusion Criteria:

* Presence of uncontrolled and/or untreated periodontal disease.
* Patients currently smoking cigarettes, cannabis, and electronic cigarettes.
* Subjects taking medications known to impact bone metabolism or have the capacity to affect wound healing. These drugs include bisphosphonates, corticosteroids, parathyroid hormone, RANKL inhibitors, past exposure to head and neck radiation, chemotherapy within the last 12 months, among others.
* Subjects with systemic diseases that impact bone metabolism and wound healing. Namely, osteoporosis, osteopenia, hyperparathyroidism, Paget's disease.
* Allergy to the graft materials.
* Pregnant subjects or individuals who self-report as attempting to become pregnant.
* Patient's unwilling to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Horizontal linear change of the buccal bone | 6 months
  Radiographic changes of bone level in mm based on cone-beam computed tomography

SECONDARY OUTCOMES:
The volumetric changes of the facial soft tissue | 6 months
  Volumetric changes in mm^3 based on intraoral digital scans
The vascular changes of the facial soft tissue | 6 months
  Vascular changes in mm^3 based on ultrasound scans
Peri-implant health, as defined by clinical attachment level. | 6 months
  Changes in clinical attachment level measurements in mm
Patient-reported morbidity, satisfaction and comfort using a visual analogue scale (VAS) | 6 months
  Difference in survey results
Clinician-reported overall treatment effectiveness | 6 months
  Scale from 1 (Poor) to 5 (Excellent)
Histological bone density | 6 months
  Histomorphometry

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Saleh, BDS, MSD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No